CLINICAL TRIAL: NCT00692250
Title: A Phase I Open Label, Randomised, Single Dose, 2-way Crossover, 2-Sequence Pharmacokinetic Study on the Interaction of Colesevelam and Ciclosporin in Healthy Volunteers
Brief Title: A Study to Assess Any Potential Interaction Between Colesevelam and Ciclosporin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CHOL00207; EudraCT 2007-003724-38
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Colesevelam hydrochloride film-coated tablets (Cholestagel)

SUMMARY:
This study is designed to assess any potential interaction between colesevelam and ciclosporin in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a body mass index (BMI) between 19 and 25 inclusive
* Medically healthy subjects with clinically normal laboratory profiles, physical exams, vital signs and ECGs.
* Give voluntary written informed consent to participate in the study

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic renal, hematologic, gastrointestinal (inclusive of dysphagia, swallowing disorders, severe gastrointestinal motility disorders), endocrine, immunologic, dermatologic, neurologic, infectious, or psychiatric disease.
* In addition, history or presence of: Alcoholism or drug abuse within the past year; OR hypersensitivity or idiosyncratic reaction to ciclosporin or other immunosuppressive agents; OR Chronic infection
* Subjects who ere tested positive at screening for HIV, HBsAg or HCV
* Subjects who received injectable corticosteroids in the 12 weeks preceding the first dose.
* Subjects who are allergic to castor oil or corn oil
* Subjects whose sitting blood pressure is less than 110/60 mmHg at screening or 100/55 mmHg before dosing
* Subjects who have used any medications or substances known to be strong inhibitors of CYP3A enzymes within 10 days prior to the first dose.
* Subjects who have used any medications or substances known to be strong inducers of CYP3A enzymes within 28 days prior to the first dose.
* Subjects who have used antibiotics within 14 days prior to the first dose.
* Subjects who have used other medication (including over-the-counter products) vitamins and herbal products within 7 days prior to the first dose.
* Subjects who have used any live attenuated vaccine within 7 days prior to the first dose or are planning to use within 14 days after the end of the study.
* Subjects who, prior to informed consent, would have donated in excess of: 500mL of blood in 14 days;1500mL of blood in 180 days; OR 2500mL of blood in 1 year.
* Subjects who have participated in another clinical trial: within a period less or equal to 2 half live (t1/2) of the previous investigational product used OR within 60 days prior to first dose.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Ciclosporin (AUC(0-t), AUC(∞) and C(max)) | 12 weeks

SECONDARY OUTCOMES:
Safety | 12
Tolerability | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- University Medical Center Groningen- Biotech Center, Groningen, Netherlands